CLINICAL TRIAL: NCT02102477
Title: Primary Radical Prostatectomy Versus Primary Radiotherapy for Locally Advanced Prostate Cancer: an Open Randomized Clinical Trial
Brief Title: Surgery Versus Radiotherapy for Locally Advanced Prostate Cancer
Acronym: SPCG-15
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olof Akre (Other)
Responsible Party: Sponsor-Investigator, Olof Akre, Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPCG-15
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic neoplasms; Locally advanced; Radiotherapy; Surgery; Mortality
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prostatectomy; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prostatectomy/Surgery (Experimental): Patients with locally advanced prostate adenocarcinoma recieves Prostatectomy/Surgery with or without adjuvant or salvage radiotherapy
  Interventions: Procedure: Prostatectomy/Surgery
- Radiotherapy with adjuvant androgen deprivation therapy (Active Comparator): Patients with locally advanced prostate adenocarcinoma treated with adjuvant androgen deprivation therapy
  Interventions: Other: Radiotherapy with adjuvant androgen deprivation therapy

INTERVENTIONS:
Procedure: Prostatectomy/Surgery — Radical prostatectomy with or without adjuvant or salvage radiotherapy
  Arms: Prostatectomy/Surgery
Other: Radiotherapy with adjuvant androgen deprivation therapy — Radiotherapy with adjuvant androgen deprivation therapy
  Arms: Radiotherapy with adjuvant androgen deprivation therapy

SUMMARY:
This prospective, open randomized phase III surgical trial seeks to study whether radical prostatectomy (with or without the combination of external radiation) improves prostate-cancer specific survival in comparison with primary radiation treatment and hormonal treatment among patients diagnosed with locally advanced (T3) prostate cancer. Untreated or conservatively treated locally advanced prostate cancer is associated with high mortality. Modern curative treatment for advanced solid malign tumors include surgery and/or radiation plus attempted chemotherapy if available to achieve both local control and elimination of potential micro metastases. Whereas there is evidence that surgery can cure localized prostate cancer, there are no clinical trials of multi-modal treatment of locally advanced prostate cancer that includes surgical removal of the prostate.

One potential advantage of adding prostatectomy to the treatment of LAPC is that removing the prostate enables a full pathological assessment of the tumor characteristics and thus a better estimation of the risk of recurrence. Surgical treatment could thus reduce the numbers needed to treat with chemotherapy and radiation, and thus improve quality of life after treatment. In addition, evidence indicate that residual cancer in the prostate occurs in 25% after radiation treatment (56) and surgical removal of the prostate may improve survival beyond what can be achieved by radiation and ADT. On the other hand, patients treated with surgery, radiation and hormones will experience side effects of all three treatment modalities and might fare better if radiotherapy plus hormones can provide oncological control without prior surgery.

A randomized clinical trial comparing two multimodal treatment regimens of which one includes a radical prostatectomy is therefore warranted.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤75, at the time of randomization
* Diagnosed histopathologically confirmed and untreated prostatic adenocarcinoma
* The general condition and mental status of patients shall permit observation in accordance with the study protocol
* Tumor stage (T, M, N):

T3 stage (as indicated by digital rectal examination or MR imaging or other validated imaging technique) T4 tumors can be included if considered resectable/treatable on MR imaging Significant extra-capsular tumor extension in biopsy (rare but acceptable for inclusion) M0 (no sign of distant metastases) confirmed by bone scan or CT or MRT of axial skeleton (at a maximum of pelvis and lumbar vertebral column) N0 stage, defined in accordance to the RECIST guidelines as no sign of macroscopic retroperitoneal lymph-node metastases >=1.5 cm (short axis) on CT scan, PET-CT, or MRT or more than one suspected lymph-node metastases Presence Gleason grade pattern 4 or 5

- Signed Informed consent

Exclusion Criteria:

* Patients with a PSA value of > 100 ng/mL
* Any medical condition that, in the opinion of the investigator, might interfere with the evaluation of the study objectives Patients with contraindications for either prostatectomy or radiotherapy to the prostate are not eligible for the study. Most contraindications for these treatments are relative, but in general, radiotherapy may be precluded among patients with:
* Anorectal disease, such as fistulae, Crohn´s disease, and ulcerative colitis
* Significant obstructive lower urinary tract symptoms
* Proximal stricture of the urethrae
* Severe neurogenic bladder dysfunction
* Enlarged prostate beyond 70-90 ml
* Previous radiotherapy to the pelvic region

On the other hand, surgery may be precluded among patients with:

* Massive local tumor progression, particularly in the apical region
* Massive abdominal obesity
* Contraindications to anesthesia

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2045-12 (Estimated)

PRIMARY OUTCOMES:
Cause specific survival | Up to 10 years
  Cause-specific survival (CSS) will be calculated as "1-cause specific mortality. Mortality and mortality causes will be ascertained from the nationwide Cause-of-Death Register. In the absence of a functioning Cause-of-Death register, an endpoint committee of at least 2 medical doctors will determine the cause of death.

SECONDARY OUTCOMES:
Metastasis free survival | Up to 10 years
  Composite endpoint of time to metastasis and survival
Quality of life - general psychological, urinary, bowel and sexual health | At 1,2,5 and 10 years after randomization
  Questionnaire-based evaluation of general psychological health, urinary health, bowel health, and sexual health.
  Questions about self Questions about quality of life in the past month (scale 1 to 7; 1=no quality, 7=the best quality) Depression and anxiety (scale 1 to 7; 1=no, 7=very) Symptom Form (EPIC-26) (scale 1 to 5; 1= no problem, 5=major problem) Questions about the urinary tract Questions about sexual function Questions about bowel function Questions about prostate cancer - diagnosis and treatment Questions about prostate cancer check-ups Questions about hormone/castration therapy and its significance Questions about pain and lymph swelling
Overall survival | Up to 10 years
  Overall survival (OS) will be calculated as "1-overall mortality. Mortality data will be ascertained through the nationwide Cause-of-Death Register.
Time to castration-resistant prostate cancer | Up to 10 years
  Ascertained at follow-up visits
Time to biochemical progression | Up to 10 years
  Ascertained at follow-up visits
Adverse events | Up to 10 years
  Ascertained at visits
Cardiovascular disease | Up to 10 years
  Data from national PcBaSe-register (https://snd.gu.se/en/catalogue/study/ext0014), a registry where the national prostate cancer registry (NPCR, www.npcr.se) has been linked to the Swedish National Cancer Register, the Cause of Death Register, the Prescribed Drug Register, the National Patient Register, and the Acute Myocardial Infarction Register, the Register of the Total Population, the Longitudinal Integration database for health insurance and labour market studies (LISA), the Multi-Generatioon Register and several other population-based registers.

OTHER OUTCOMES:
Health-care consumption | Annually up to 10 years
  Annual Defined Daily Dose (DDD) of analgesics, prescription databases
Health-care consumption | Annually up to 10 years
  Annual number of days of hospitalization from patient registers

CONTACTS AND LOCATIONS:
Overall Officials: Johan Stranne, M.D ass prof, Principal Investigator — Sahlgrenska University Hospital, Department of Urology, SE- 413 45 Gothenburg; Camilla Thellenberg Karlsson, MD, PhD, Principal Investigator — Umeå University Hospital, Department of Radiation Science, SE-901 87 Umeå Sweden; Eva M Johansson, R.N PhD, Principal Investigator — Karolinska Institute, Nobelsväg, SE- 171 77 Solna, Sweden; Gunnar Steineck, M.D Prof, Principal Investigator — Karolinska Institute, Nobelsväg, SE-171 77 Solna, Sweden; Klaus Brasso, M.D, Principal Investigator — Rigshospitalet, department Urology, DK-2001-Copenhagen, Denmark; Peter M Meidahl Petersen, M.D ass prof, Principal Investigator — Rigshospitalet, Region h, Department of Oncology, Blegdamsvej 9, DK- 2001, Copenhagen, Denmark; Bjørn Brennhovd, M.D ass.prof, Principal Investigator — Oslo University Hospital, Department of Urology, P.O Box 4950 Nydalen, N-0424, Oslo Norway; Wolfgang Lilleby, M.D ass.prof, Principal Investigator — Oslo University Hospital, Department of Radiation Therapy, P.O Box 4950, N-0424, Nydalen Oslo, Norway; Antti Rannikko, M.D ass.prof, Principal Investigator — Helsinki University Central Hospital, Department Urology,Stenbäckinkatu 9, FIN-00290 Helsinki , Finland; Mauri Kouri, M.D PhD, Principal Investigator — Helsinki University Central Hospital, Department Urology,Stenbäckinkatu 9, FIN-00290 Helsinki , Finland; Tuomas Mirtti, M.D PhD, Principal Investigator — Helsinki University Central Hospital, Department Urology,Stenbäckinkatu 9, FIN-00290 Helsinki , Finland
Locations (30):
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Region h, Department Oncology, Copenhagen
  - Rigshopsitalet Department urology, Copenhagen
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense
- Finland (3):
  - Helsinki University Hospital, Department of Urology, Helsinki
  - Tampere University Hospital, Pihlajalinna Koskiklinikka, Tampere
  - Turku University Hospital, Turku
- Norway (5):
  - Sørlandet Hospital, Kristiansand
  - Oslo University Hospital, Department of radiation Therapy, Oslo
  - Oslo University Hospital, Department Urology, Oslo
  - University Hospital of North Norway, Tromsø
  - St. Olavs Hospital, Trondheim
- Sweden (16):
  - Falu Lasarett, Falun
  - Sahlgrenska University Hospital, Gothenburg
  - Helsingborgs Lasarett, Helsingborg
  - Länssjukhuset Ryhov, Jönköping
  - Kirurgkliniken, Blekingesjukhuset, Karlskrona
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Malmo
  - Vrinevis Hospital, Norrköping
  - Östersund Hospital, Östersund
  - Karolinska University Hospital, Stockholm
  - Capio St Göran Hospital, Stockholm
  - Sundvalls Hospital, Sundsvall
  - Umeå University Hospital, Umeå
  - Uppsala Akademiska Hospital, Uppsala
  - Centrallasarettet, Vaxjo
  - Centrallasarettet Växjö Hospital, Vaxjo

IPD SHARING:
Plan to Share IPD: Yes